CLINICAL TRIAL: NCT06002893
Title: The Antihypercholestrolemic Pharmacological Effect of a Combined Supplement of Amla Fruit, Walnut Leaves, Red Yeast Rice, and Olive Fruit Extracts Leads to Improvement in Circulatory Levels of LDL-C and Remnant Cholesterol
Brief Title: The Antihypercholestrolemic Effect of a Combined Nutritional Supplementation of Standardized Extracts of Amla, Walnut, Red Yeast Rice and Olive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK/08.08.2023/01
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Cholesfytol NG®) supplement treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cholesfytol NG®) supplement (Experimental): Patients will receive a single oral dose of 2 tablets a day of Cholesfytol NG®) supplement for 2-months.
  Interventions: Dietary Supplement: Cholesfytol NG®) supplement

INTERVENTIONS:
Dietary Supplement: Cholesfytol NG®) supplement — General Practitioner (GP) prescribed oral Cholesfytol NG®) supplement

SUMMARY:
Nutraceutical lipid-lowering interventions are becoming increasingly popular, particularly among patients who are intolerant or refractory to prescription statins, or who desire alternative non-conventional pharmacological treatment to manage their dyslipidaemia, whether they previously experienced statin intolerance or not. A growing body of preclinical and clinical evidence suggest that the amla (Emblica officinalis) red yeast rice (RYR), olive and walnut leaf extracts posses consideable hpolipidaemic pharmacological effects.

DETAILED DESCRIPTION:
The present exploratory study aimed to assess the safety, efficacy, and patient's satisfaction of a combined supplementation of amla, red yeast rice, olive, and walnut leaf extracts (Cholesfytol NG®) on total cholesterol (TC), low-density lipoprotein - cholesterol (LDL-C), high-density lipoprotein - cholesterol (HDL-C), non-high-density lipoprotein - cholesterol (non-HDL-C), remnant cholesterol (RC) and triglycerides (TG) in hyperlipidaemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Both male or female
* Blood total cholesterol (TC) level ≥ 200 mg/dL
* Blood low-density lipoprotein cholesterol (LDL-C) level ≥ 130 mg/dL
* With or without myalgia and/or diabetes
* No prior treatment of cholesterol-lowering agents and/or patients whose cholesterol- lowering treatment did not allow them to reach LDL-C target
* Patients who had stopped their cholesterol-lowering treatment because of side effects including myalgia

Exclusion Criteria:

* Pregnant nor breastfeeding patients

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in blood lipid profile | 2-months
  Decrease in blood total cholesterol (TC) concentration
Change in blood lipid profile | 2-months
  Decrease in blood low-density lipoprotein - cholesterol (LDL-C) concentration
Change in blood lipid profile | 2-months
  Decrease in blood triglycerides (TG) concentration
Change in blood lipid profile | 2-months
  Decrease in blood non-high density lipoprotein - cholesterol (non-HDL-C) concentration
Decrease in blood lipid profile | 2-months
  Change in blood remnant cholesterol (RC) concentration

SECONDARY OUTCOMES:
Rate of side effects | 2-months
  Number of patients reporting myalgia

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires St-Luc and Institut de Recherche Expérimentale et Clinique (IREC), KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hermans MP, Dierckxsens Y, Janssens I, Seidel L, Albert A, Ahn SA, Rousseau MF, Khan A. The antihyperlipidemic effect of a combined supplement of standardized dry extracts of amla (Emblica officinalis), walnut (Juglans regia), olive (Olea europaea) and red yeast rice (Monascus purpureus) powder: Reduction in circulatory low-density lipoprotein-cholesterol (LDL-C) and remnant cholesterol (RC) levels in patients with hypercholesterolemia. Front Pharmacol. 2023 Nov 27;14:1280234. doi: 10.3389/fphar.2023.1280234. eCollection 2023. PMID 38089061